CLINICAL TRIAL: NCT06554327
Title: Fast Multiplex PCR of Bronchoalveolar Lavage for Antibiotic Stewardship in Ventilator Associated Pneumonia. A Multicenter, Randomized Controlled Study
Brief Title: Ventilator Associated Pneumonia Multiplex PCR for Anti-Infective Regimens
Acronym: VAMPAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR24072
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator associated pneumonia; Intensive care unit; Empirical antimicrobial therapy; Multiplex PCR; Diagnosis; Antibiotic stewardship; Bronchoalveolar lavage
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Disease | interventions — Multiplex Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Device: Multiplex PCR
- control group (Active Comparator)
  Interventions: Device: Multiplex PCR

INTERVENTIONS:
Device: Multiplex PCR — In the intervention group (Multiplex PCR performed and results communicated to the clinician), bronchoalveolar lavage will be examined directly after Gram staining by the laboratory, followed by quantitative culture. A multiplex PCR will be performed.

SUMMARY:
Ventilator-associated pneumonia (VAP) remains one of the main nosocomial infections acquired in the intensive care unit (ICU). VAP is pneumonia occurring 48 hours after intubation. Today, bronchoalveolar lavage (BAL) is used for microbiological diagnosis, with bacterial culture and antibiotic susceptibility results within 48 to 72 hours. Multiplex PCR can detect DNA of a number of bacteriae, as well as the presence of resistance genes. However, its clinical value in the ICU remains to be demonstrated. We think that the use of multiplex PCR with a panel adapted to the microbiology of VAP, could be an interesting method for clinicians in ICU.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) remains one of the main nosocomial infections acquired in the intensive care unit (ICU). VAP is pneumonia occurring 48 hours after intubation. Today, bronchoalveolar lavage (BAL) is used for microbiological diagnosis, with bacterial culture and antibiotic susceptibility results within 48 to 72 hours. Multiplex PCR can detect the bacterial DNA of a number of bacteria, as well as the presence of resistance genes. However, its clinical value in the ICU remains to be demonstrated. We think that the use of multiplex PCR with a panel adapted to the microbiology of VAP, could be an interesting method for clinicians in ICU.

The aim of our study is to compare the percentage of appropriate empirical antibiotic therapy in the group benefiting from multiplex PCR on BAL prior to bacterial culture results compared to control group (bacterial culture alone=usual management) in patients with culture-confirmed VAP.

This is a multicenter, randomized, controlled, French study conducted in 8 university intensive care units (2 surgical units, 6 medical units) in the Grand-Est region of France. The multiplex PCR tested here is BioFire's FilmArray Pneumonia Panel Plus. It is performed solely on per-fibroscopic bronchoalveolar lavage (BAL) fluids in cases of suspected VAP.

ELIGIBILITY:
inclusion criteria :

* Adult patients, hospitalized in intensive care unit
* on mechanical ventilation for at least 48 hours
* Suspected VAP
* With an indication for bronchoalveolar lavage (BAL)

exclusion criteria :

* Patients under legal protection or without social security coverage
* Pregnant women
* Previous episode of VAP during the same hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2026-09-06 (Estimated); Study Completion 2026-10-06 (Estimated)

PRIMARY OUTCOMES:
The percentage of appropriate empirical antibiotic therapy in cases of culture-confirmed VAP, according to the diagnostic method used (multiplex PCR or not). | Day 14
  The appropriate antibiotic is one that is effective against the diagnosed pathogen and has the narrowest possible antibiotic spectrum.

SECONDARY OUTCOMES:
The percentage of effective antibiotic treatment for the identified germ in each group. | Day 14
  The effective antibiotic is one that is effective against the diagnosed pathogen.
Duration of inappropriate antibiotic therapy (in hours) in each group | Day 14
  An inappropriate antibiotic is one that is not active according to the in vitro antibiogram of the identified pathogen, or whose spectrum is too broad for the resistance profile of the identified pathogen.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

IPD SHARING:
Plan to Share IPD: No